CLINICAL TRIAL: NCT06453395
Title: PPIO-009 Tumor Regression Grade and Prognosis Analysis of Esophageal Cancer in Different Tumor Location After Neoadjuvant Immunotherapy
Brief Title: PPIO-009 Tumor Regression Grade and Tumor Location in Esophageal Cancer
Status: Completed | Type: Observational
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, WEI GUO, chief physician, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Other Study IDs: NO:2023(289)
Record Dates: First submitted 2024-06-04; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Tumor Regression Grade

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- upper thoracic case: Cervical esophagus to lower border of the azygos vein
  Interventions: Other: Patients were grouped according to tumor location
- Middle thoracic case: Cervical esophagus to lower border of the azygos vein
  Interventions: Other: Patients were grouped according to tumor location
- Lower thoracic case: Lower border of the inferior pulmonary vein to the stomach, including the esophagogastric junction
  Interventions: Other: Patients were grouped according to tumor location

INTERVENTIONS:
Other: Patients were grouped according to tumor location — Patients were grouped according to tumor location

SUMMARY:
At present, the evaluation of the effect of neoadjuvant chemoradiotherapy combined with immunotherapy for locally advanced esophageal cancer is mainly based on postoperative pathology, among which, the pathological assessment of tumor regression grade (TRG) and TNM staging are the basis for the routine pathological diagnosis of esophageal cancer, and the College of American Pathologists divides the TRG after neoadjuvant therapy to esophageal cancer into four grades: 0, 1, 2, and 3.The residual primary tumor in the resection specimen following neoadjuvant therapy is associated with shorter overall survival. Therefore ，the prediction of TRG after neoadjuvant therapy is vital for patients. We aim to seek to identify factors associated with TRG system as defined by the NCCN.

DETAILED DESCRIPTION:
Oesophageal cancer is the eighth most common cancer globally (934,870 new cases) and the sixth most common cause of cancer death (287,270 new deaths).The incidence, prevalence, and histological type of oesophageal cancer vary geographically , with about 75% of cases occurring in Asia, with China having the highest share, accounting for about 50% of the total cases and cancer-specific deaths. According to the National Bureau of Statistics of China, Statistics 2022, there were 252,500 cases of oesophageal cancer and 193,900 deaths in China in 2016, making oesophageal cancer the sixth most common cancer and the fifth leading cause of cancer death in China . The etiology of the two most common histological subtypes (esophageal squamous cell carcinoma [ESCC] and adenocarcinoma) varies widely. In the West, heavy alcohol consumption and smoking and their synergistic effects are the main risk factors for ESCC . However, in low-income countries, such as parts of Asia and sub-Saharan Africa, the main risk factors for ESCC, which typically accounts for more than 90% of all oesophageal cancer cases, have not been elucidated.

Preclinical studies have shown that the PD-1/PD-L1 axis can be activated early in solid tumours , and a durable protective effect may occur with preoperative induction of the immune response. Considering the dramatic decrease in tumour antigens after surgical resection and the removal of intact blood vessels and lymph nodes delivering the drug may affect the immunotherapeutic efficacy, the use of immunotherapy preoperatively may be more effective. Several phase 1/2 and phase 2 studies have shown a manageable safety profile and preliminary demonstration of efficacy when PD-1/PD-L1 inhibitors were added to perioperative therapy in resectable EC subjects. PD-1 inhibitors have demonstrated significant benefit in both second-line therapy and first-line therapy. Given the evidence of antitumour activity of immunotherapy in patients with ESCC and the continuing need to improve survival and reduce recurrence rates in resectable oesophageal cancer, a number of studies exploring the antitumour activity of immunotherapy in the treatment of resectable disease have tentatively shown promise as a neoadjuvant therapy.

Currently, after patients receive neoadjuvant therapy, tumour cell regression can occur with a variety of histological changes, such as tumour cell necrosis and apoptosis, fibrous tissue proliferation, inflammatory cell infiltration, foam cell aggregation, cell-free mucus production and formation of mucus pools, as well as calcified foci formation. However, not all tumours produce the above regression reactions after treatment, fibrohistiocytosis and inflammatory cell infiltration are the most common histological regression changes, and in order to assess the clinical therapeutic efficacy of the tumour, tumour regression needs to be graded quantitatively.TRG is a quantitative analysis of the pathology of tumours resected after neoadjuvant chemotherapy to clarify the therapeutic efficacy of chemotherapy or targeted drugs on tumours and to predict the patient's postoperative recurrence and metastasis. Metastasis. It was firstly used to assess the efficacy of oesophageal cancer after concurrent radiotherapy; and then gradually used to assess the efficacy of oesophageal cancer. The current assessment of post-radiotherapy samples is mainly based on the proportion of residual tumour components and fibrosis to grade pathological regression. Currently, the main methods for TRG scoring after neoadjuvant radiotherapy include NCCN, AJCC and other standards.

Currently, based on the data of pre-surgical clinical studies, the remission rate after neoadjuvant therapy varies in different oesophageal segments, which may indicate that the difference in blood supply of oesophageal cancer in different segments affects the blood drug concentration, leading to different clinical outcomes in patients with oesophageal cancer in different segments. In order to better treat patients in different segments, it is necessary to establish a prediction model based on the clinical data of patients in different oesophageal segments for better clinical decision-making.

ELIGIBILITY:
Inclusion Criteria:

* 1. Clinical diagnosis of Esophageal Squamous Cell Carcinoma 2. patients with clinical TNM (cTNM) stage II-IVA ESCC 3. patients with Neoadjuvant Immunochemotherapy before esophagectomy

Exclusion Criteria:

* 1. nonradical resection (R1 or R2) 2. combined with other anticancer therapies (radiotherapy or Targeted drugs) 3. incomplete data or missing follow-up time 4. concurrent or previous presence of malignancies at other sites

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: From January 1, 2019 to October 1, 2023 thoracoscopic esophagectomies for ESCC of the thoracic esophagus were performed in the Department of Thoracic Surgery, Daping Hospital, Army Medical University (Chongqing, China)
Sampling Method: Non-Probability Sample
Enrollment: 248 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-06-04 (Actual)

PRIMARY OUTCOMES:
Tumor regression grade | up to 1 weeks
  Tumor regression grade was defined by NCCN/CAP system. The grading ranges from 0 to 3. TRG is scored as follows: grade 0-No viabal cancer cell (including lymph nodes), grade 1-single cells or small groups of cancer cells, grade 2-single cells or rare small groups of cancer cells, and grade 3-extensive residual cancer with no evident tumor regression.

SECONDARY OUTCOMES:
Disease-free survival | About 2 years postoperatively
  Disease-free survival (DFS) was defined as the time from the date of surgery to recurrence, metastasis, and death from any cause.
Overall survival | About 2 years postoperatively
  Overall survival (OS) was defined as the time from the date of surgery to death from any cause or last follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Army Medical Center of the People's Liberation Army, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No